CLINICAL TRIAL: NCT06809764
Title: Clinical Effectiveness and Safety of Trastuzumab Deruxtecan in Chinese Patients With HER2 Mutant Metastatic Non-small Cell Lung Cancer: a Prospective, Observational Study (RERUN)
Brief Title: Clinical Effectiveness and Safety of Trastuzumab Deruxtecan (T-DXd) in Chinese Patients With HER2m NSCLC (RERUN)
Acronym: RERUN
Status: Recruiting | Type: Observational
Sponsor: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Other Study IDs: DS8201-0079-NIS-MA
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Locally advanced or metastatic NSCLC; HER2 mutations; T-DXd
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NSCLC patients with HER2 mutations: Patients with NSCLC with HER2 mutations who receive T-DXd based on physician's decisions will be enrolled.
  Interventions: Other: No drug

INTERVENTIONS:
Other: No drug — This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol; however, participants on T-DXd will be enrolled in this study.

SUMMARY:
Trastuzumab deruxtecan (T-DXd) is an approved therapy for non-small cell lung cancer (NSCLC) in China. Despite the clinical trial evidence, there is no real-world data of T-DXd used in Chinese lung cancer patients with HER2 mutations.

This real world, prospective study will assess the effectiveness and safety of T-DXd in patients with locally advanced or metastatic, HER2 mutation-positive NSCLC in real-world setting.

DETAILED DESCRIPTION:
T-DXd is an approved therapy in China for locally advanced or metastatic NSCLC patients with human epidermal growth factor receptor 2 mutations (HER2m). In previous clinical trials, T-DXd demonstrated efficacy and manageable safety profiles in the ≥ second-line setting for NSCLC harboring HER2m. However, patient populations are more diverse in routine practice and no real-world data of T-DXd used in Chinese lung cancer patients with HER2 mutations exist.

This study will assess the effectiveness of ≥ second-line treatment of T-DXd in real-world setting as the primary objective. Secondary objectives will further assess the effectiveness and overall survival of ≥ second-line treatment of T-DXd in real-world setting as well as evaluate the safety and tolerability of any-line treatment of T-DXd in real-world setting. This is an non-interventional, observational study. No drug will be provided or administered as part of this protocol; however, participants on T-DXd will be enrolled in this study.

ELIGIBILITY:
The key inclusion criteria for this study are:

1. Age ≥18 years at signing informed consent form (ICF).
2. Pathologically documented unresectable and/or metastatic non-squamous NSCLC.
3. Documented any known activating HER2 mutation.
4. Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2.
5. Patients who receive T-DXd based on physicians' discretion (Newly received or just have started the first dose no longer than 2 months before enrollment).

The key exclusion criteria for this study are:

1. Previously treated with HER2-targeted/directed therapies, including:

   * tyrosine kinase inhibitors [TKIs] targeting HER2 mutations, except for pan-HER class TKIs.
   * an ADC, containing a chemotherapeutic agent targeting topoisomerase I
2. Has spinal cord compression or clinically active CNS metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms.
3. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension active bleeding diatheses, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC patients with HER2 mutations who receive T-DXd based on physicians' discretion will be enrolled from about 30 sites in China.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) by Investigator Assessment in Real-world Setting (rwPFS) | Baseline up to approximatley 2 years
  rwPFS is defined as the time from the initiated date of ≥ second-line treatment of T-DXd until disease progression or death by investigator report as recorded in the electronic case report forms (eCRF).

SECONDARY OUTCOMES:
Time to Treatment Discontinuation or Death (TTD) | Baseline up to approximately 2 years
  TTD is defined as the time from the initiated date of ≥ second-line treatment of T-DXd to the date of treatment discontinuation or death from any cause.
Best Overall Response Rate (BORR) | Baseline up to approximately 2 years
  BORR is defined as the percentage of patients with complete response (CR) or partial response (PR) as assessed by investigator for ≥ second-line treatment of T-DXd. Based on RECIST guidelines, CR was defined as a disappearance of all target lesions and PR was defined as at least a 30% decrease in the sum of diameters of target lesions.
Overall Survival | Baseline up to approximately 2 years
  Overall survival is defined as the time from the initiated date of ≥ second-line treatment of T-DXd until death due to any cause.
Number of Patients Reporting Treatment-related Adverse Events (TRAEs), Adverse Events of Special Interests (AESIs), and AEs Leading to Dose Interruption, Reduction, Discontinuation | Baseline up to approximately 2 years
  TRAEs, AESIs and AEs leading to dose interruption, reduction, discontinuation will be graded by the investigators using National Cancer Institute (NCI) common terminology criteria for adverse events (CTCAE) version 5.0 and coded using the medical dictionary for regulatory activities (MedDRA).

CONTACTS AND LOCATIONS:
Overall Officials: Project Manager, Study Director — Daiichi Sankyo Co., Ltd.
Locations (23):
- China (23):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing
  - Peking University International Hospital, Beijing
  - Beijing Cancer Hospital, Beijing
  - Hunan Second People's Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou
  - Zhejiang Cancer Hospital, Hangzhou
  - Anhui Provincial Cancer Hospital, Hefei
  - First Affiliated Hospital of Shandong First Medical University, Jinan
  - Cancer Hospital of Shandong First Medical University, Jinan
  - The First Affiliated Hospital of Jinzhou Medical University, Jinzhou
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Guangxi Medical University Cancer Hospital, Nanning
  - Ruijin Hospital, Shanghai Jiaotong University School Of Medicine, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - Cancer Hospital Chinese Academy of Medical Sciences, Shenzhen Center, Shenzhen
  - The Fourth Hospital of Hebei Medical University, Shijiazhuang
  - Shangxi Provincial Cancer Hospital, Taiyuan
  - The First Affiliated Hospital of Xiamen University, Xiamen
  - Henan Cancer Hospital, Zhengzhou
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou

IPD SHARING:
Plan to Share IPD: No